CLINICAL TRIAL: NCT00482820
Title: A Clinical Research Studying a Method of Intervention for Children Diagnosed With Anxiety Disorder: Attentional Bias Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, alan apter, Director, Feinberg Child Study Center and Department of Psychiatry, Schneider's Children's Medical Center of Israel, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 4373
Record Dates: First submitted 2007-06-04; First posted 2007-06-05 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Anxiety
Keywords: anxiety; attention-biases; children
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- 1 (Experimental): attention training away from threat
  Interventions: Behavioral: attention-bias training
- 2 (Placebo Comparator): placebo attention training
  Interventions: Behavioral: attention-bias training

INTERVENTIONS:
Behavioral: attention-bias training — one group recive an attention training away from threat. The second group, the controll group, recive a placebo training

SUMMARY:
Studies show that children with high levels of anxiety tend to pay more attention to threatening stimulus in the environment. They tend to attend to these stimuli and have difficulty to disengage from them. These attention biases enhance and maintain the level of anxiety. The aim of this study is to test a method of therapeutically intervention which focuses on shifting these attentional biases, with the use of a computer game which was designed to train the child to focus his/her attention away from the threatening stimuli and to focus on natural or positive stimuli. We will recruit 160 children with ongoing anxiety disorders who seek treatment. We will first assess threat-related attention bias and anxiety symptoms using structured psychiatric interviews and questionnaires. We will then randomly assign these children to one of four conditions: training to avoid threatening stimuli and attend to neutral stimuli; control placebo-training for threat-neutral stimuli; training to attend to positive stimuli and avoid neutral stimuli; and, control placebo-training for positive-neutral stimuli. Upon completion of training we will again assess attention bias and anxiety.

Two sets of predictions will be tested, one set concerns the effects of training on attention, and the other concerns the effects of training on anxiety. In terms of training effects on attention, we hypothesize that children with anxiety disorders can be trained to either avoid threat or attend to positive stimuli. In terms of training effects on anxiety symptoms, we hypothesize that the experimental training sessions will produce greater reduction in symptoms of anxiety than the placebo-control training sessions.

ELIGIBILITY:
Inclusion Criteria:

* Children with Clinical diagnosis of Generalized Anxiety Disorder (GAD), Social Phobia (SP), or Separation Anxiety Disorder (SAD).

Exclusion Criteria:

* Children with the diagnoses of OCD, specific phobia, and PTSD in the absence of comorbid GAD, SP, or SAD.
* Other exclusion criteria include ongoing major depressive disorder, and use of psychotropic medication.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2007-07; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
anxiety questionnaire - that are specified in the protocol. mood scale- as described in the protocol attention bias scores- as described in the protocol | 2-4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bar-Haim Yair, Phd, Study Director — Tel-aviv university; and schnider children's medical center of isreal

REFERENCES:
- [Derived] Eldar S, Apter A, Lotan D, Edgar KP, Naim R, Fox NA, Pine DS, Bar-Haim Y. Attention bias modification treatment for pediatric anxiety disorders: a randomized controlled trial. Am J Psychiatry. 2012 Feb;169(2):213-20. doi: 10.1176/appi.ajp.2011.11060886. PMID 22423353